CLINICAL TRIAL: NCT00296894
Title: TNF-Blockade for the Treatment of Erosive Osteoarthritis (OA) of Interphalangeal Finger Joints: Randomized, Double Blind, Placebo-Controlled Cross-Over Study to Evaluate the Efficacy of Adalimumab 40 mg SC Every Other Week in Patients With Erosive Osteoarthritis of the Interphalangeal Finger Joints
Brief Title: Study to Evaluate the Efficacy of Adalimumab in Patients With Erosive Osteoarthritis of the Interphalangeal Finger Joints
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Gust Verbruggen, University Hospital Ghent
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2006/072
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Erosive Osteo-Arthritis
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Drug - adalimimab sc
  Interventions: Drug: Adalimumab (40 mg sc every other week)
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adalimumab (40 mg sc every other week) — Adalimumab (40 mg sc every other week)
  Arms: 1
Drug: Placebo — Placebo
  Arms: 2

SUMMARY:
Patients will be randomized into two groups (1/1) during one year:

* 40 mg adalimumab subcutaneously (sc) every other week
* placebo

The effect on x-rays and clinical parameters will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Clear erosive image on x-ray of at least one interphalangeal finger joint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-05; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Evaluation of x-rays
Evaluation of clinical parameters (pain, daily functioning, etc.)

CONTACTS AND LOCATIONS:
Overall Officials: Gust Verbruggen, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be